CLINICAL TRIAL: NCT02514005
Title: Effectiveness of Manual Therapy and Dry Needling in Nonspecific Patellofemoral Syndrome.
Brief Title: Manual Therapy and Dry Needling in Patellofemoral Syndrome
Acronym: MTPSSFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Dr, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ID007
Record Dates: First submitted 2015-07-27; First posted 2015-08-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Patellofemoral Syndrome
Keywords: Trigger points; Manual therapy; Patellofemoral syndrome; Dry needling
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Musculoskeletal Manipulations; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual therapy (Active Comparator): Overall bilateral manipulation (L5-S1-SI), Hip joint gapping, Stretching the hip rotators with hip and knee flexion, Femorotibial Gapping, Decompression of connective tissue of the patellofemoral region, Internal and external joint line opening in laterality, Mobilization of the base of the fibula, Tibiofibular-talus gapping, and Muscle strengthening.
  Interventions: Other: Manual therapy
- Manual therapy and Dry needling (Experimental): Dry needling is performed in the MTrPs of the vastus lateralis and vastus medialis muscles of the quadriceps.
  Interventions: Other: Manual therapy; Device: Dry needling

INTERVENTIONS:
Other: Manual therapy — - Manual Therapy. Study treatment consists of a comprehensive joint treatment of the lumbar region and the lower limbs that are related to the biomechanics of the knee. In this way, the aim is to globally balance the possible dysfunctions that may exist in the lower lumbar region and sacroiliac joint, hip, knee and ankle.
Device: Dry needling — * Manual therapy. Study treatment consists of a comprehensive joint treatment of the lumbar region and the lower limbs that are related to the biomechanics of the knee. In this way, the aim is to globally balance the possible dysfunctions that may exist in the lower lumbar region and sacroiliac joint, hip, knee and ankle.
  * Dry needling (DN). Dry needling is performed in the MTrPs of the vastus lateralis and vastus medialis muscles of the quadriceps.
  Arms: Manual therapy and Dry needling

SUMMARY:
It is a randomized clinical trial comparing two treatments in patients affected by the patellofemoral syndrome (PFS). Our aim was to investigate the effectiveness of inclusion of trigger point dry needling into the management of idividuals with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Patients The sample involved patients diagnosed with nonspecific patellofemoral syndrome. The treatment is carried out at the School of Physiotherapy (University of Valencia).

The study comprises patients with nonspecific patellofemoral syndrome. Patients excluded from the study are those with osteoarthritis, recent injuries, ligament injuries, meniscal lesions, previous injury and / or treatments lasting for a period of 6 months prior to the study.

Study design It is a single-blind randomized controlled study. 3 sessions are conducted with 7-day intervals and 15 days for the last intervention and follow-up at 3 months after treatment ended. Each session lasts approximately 30 minutes.

The sample was divided into two groups:

* Control group with manual therapy and strengthening exercises for the quadriceps and hamstrings.
* Experimental group which receives manual therapy and strengthening exercises for the quadriceps and hamstrings combined with dry needling treatment (DN) in myofascial trigger points (MTrP) of vastus medialis and vastus lateralis of the quadriceps muscle and strengthening exercises for the quadriceps and hamstrings.

Intervention Study treatment consists of a comprehensive joint treatment of the lumbar region and the lower limbs that are related to the biomechanics of the knee. In this way, the aim is to globally balance the possible dysfunctions that may exist in the lower lumbar region and sacroiliac joint, hip, knee and ankle.

Assessment

The initial assessment is a clinical interview with the characteristics of the patellofemoral syndrome for the month prior to the study and for this, the following assessment instruments are used:

* Intensity knee pain before the treatment is evaluated after treatment and monitoring.
* KOOS (Knee Injury and Osteoarthritis Outcome Score). It assesses five dimensions: pain, symptoms, activities of daily living, sport and recreational activity and quality of life related to the knee. To evaluate osteoarthritis in older patients, the 24 WOMAC questions are included.
* KSS (Knee Society Score). It is the modified scale of the American Knee Society. It makes it possible to separate the purely functional aspects of the knee joint, knee score, from those related to the patient's ability to walk and climb stairs, functional score.

It includes three main parameters (pain, stability and range of motion) and other parameters (contraction of flexion, loss of extension and alignment) considered as deductions to score of the former, possibly presenting some interobserver variation.

-IKDC (International Knee Documentation - Committee). It is an instrument to assess symptoms, function, and sport activity applicable to a variety of conditions of the knee. Validated for a variety of knee conditions including ligament, meniscal and articular cartilage injuries and also for osteoarthritis and patellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 60 years.
* Patients diagnosed with nonspecific patellofemoral syndrome. Positive sign in patellofemoral gliding test; Negetive McMurry test; Full knee range of motion; Anterior knee pain, related to prolonged sitting, climbing stairs, and descending stairs; No relevant patellofemoral degenerative changes on imaging; No history of knee trauma.

Exclusion Criteria:

* Patients excluded from the study are those with osteoarthritis, recent injuries, ligament injuries, meniscal lesions, previous injury and / or treatments lasting for a period of 6 months prior to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | up to 3 months follow up
  Intensity patellofemoral pain before the treatment is evaluated after treatment and monitoring. The pain scale was removed by the KOOS scale (Knee Injury and Osteoarthritis Outcome Score): Pain levels were assessed: absent, mild or occasional pain climbing stairs, while driving, occasional moderate, moderately severe, severe. Being 0 to 50 points = severe pain (no pain).

SECONDARY OUTCOMES:
IKDC (International Knee Documentation - Committee). | up to 3 months follow up
  It is an instrument to assess symptoms, function, and sport activity applicable to a variety of conditions of the knee. Validated for a variety of knee conditions including ligament, meniscal and articular cartilage injuries and also for osteoarthritis and patellofemoral pain.
KSS (Knee Society Score). | up to 3 months follow up
  It is the modified scale of the American Knee Society. It makes it possible to separate the purely functional aspects of the knee joint, knee score, from those related to the patient's ability to walk and climb stairs, functional score.
  It includes three main parameters (pain, stability and range of motion) and other parameters (contraction of flexion, loss of extension and alignment) considered as deductions to score of the former, possibly presenting some interobserver variation.
KOOS (Knee Injury and Osteoarthritis Outcome Score). | up to 3 months follow up
  It assesses five dimensions: pain, symptoms, activities of daily living, sport and recreational activity and quality of life related to the knee. To evaluate osteoarthritis in older patients, the 24 WOMAC questions are included.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma gemma.espi@uv.es, PhD, Principal Investigator — Department Physiotherapy. University of Valencia
Locations (1):
- Gemma V. Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Espi-Lopez GV, Serra-Ano P, Vicent-Ferrando J, Sanchez-Moreno-Giner M, Arias-Buria JL, Cleland J, Fernandez-de-Las-Penas C. Effectiveness of Inclusion of Dry Needling in a Multimodal Therapy Program for Patellofemoral Pain: A Randomized Parallel-Group Trial. J Orthop Sports Phys Ther. 2017 Jun;47(6):392-401. doi: 10.2519/jospt.2017.7389. Epub 2017 May 13. PMID 28504067